CLINICAL TRIAL: NCT04303429
Title: Adjuvant Chemotherapy Versus Observation in Stage II Colon Cancer Patients With High-Risk Factors and High-Immunoscore®
Brief Title: Adjuvant Chemotherapy in High Risk Stage II Colon Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Qi Li, Executive director of cancer center, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IMCC
Record Dates: First submitted 2020-03-05; First posted 2020-03-11 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2019-11

CONDITIONS: Stage II Colon Cancer; Adjuvant Chemotherapy
Keywords: Stage II colon cancer; Adjuvant Chemotherapy; High-Risk factors; High-Immunoscore®
MeSH Terms: conditions — Colonic Neoplasms | interventions — Folfox protocol

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- observation group (No Intervention): Patients enrolled in the observation group will not receive any chemotherapy drugs
- adjuvant chemotherapy group (Experimental): Patients enrolled in the chemotherapy group will receive postoperative chemotherapy (investigator's choice) for 3 months or 6 months.
  Interventions: Drug: FOLFOX/XELOX/Capecitabine

INTERVENTIONS:
Drug: FOLFOX/XELOX/Capecitabine — Patients enrolled in the chemotherapy group will receive postoperative chemotherapy (investigator's choice) for 3 months or 6 months.
  Arms: adjuvant chemotherapy group

SUMMARY:
* Benefit of adjuvant chemotherapy after curative surgery for stage II Colon Cancer is still debated. Several high-risk features may help to stratify stage II cancer patients into groups that will truly benefit from adjuvant chemotherapy. However, those factors are rather subjective, and no specific trial has been designed to answer the high-risk stage II colon cancer question directly.
* Immunoscore® Colon, an in vitro diagnostic test, which quantifies the density of CD3+ and CD8+ T lymphocyte populations in the center the tumor (CT) and its invasive margin (IM) using immunohistochemistry and automated image analysis. Immunoscore® has been extensively validated as a prognostic biomarker in early stage CC patients. This unique diagnostic assay measuring host immune response at the tumor site may inform the decision to administer adjuvant chemotherapy in resected Stage II and III CC patients.
* This randomized trial is studying how observation compares to adjuvant chemotherapy (investigator's choice) in stage II colon cancer patients with high-risk features and High-Immunoscore®. The trial would represent a unique opportunity to classify stage II CC patients based on their tumor microenvironment with the aim to provide efficient patient stratification to improve clinical care.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old
2. Pathologically confirmed adenocarcinoma of the colon
3. Complete resection of the primary tumor without gross or microscopic evidence of residual disease
4. Histologically proven stage II: T3-T4 N0
5. At least one of the following factors:T4 staging,Number of examined lymph nodes < 12,poor differentiation (except MSI-H),LVI or PNI,tumor perforation or occlusion
6. Treatment within 7 weeks following surgery
7. ECOG PS 0-1
8. No prior chemo, immuno or radiotherapy
9. Patients must read, agree to, and sign a statement of Informed Consent prior to participation in this study.

Exclusion criteria

1. Have a birth plan during the clinical trial;
2. Severe cardiovascular diseases such as cerebrovascular accidents occurring within 6 months, myocardial infarction, hypertension that cannot be controlled after drug intervention, unstable angina pectoris, heart failure (NYHA 2-4), and arrhythmia requiring drugs Intervention;
3. Dementia, mental state changes or any mental illness that may interfere with understanding or making informed consent or completing a questionnaire;
4. Subjects with ≥1 peripheral neuropathy according to CTCAE V version 4.03;
5. Allergy or hypersensitivity history of the drug or drug ingredient used in this test;
6. Excluding other malignant tumors, cured basal cell carcinoma of the skin or squamous cell carcinoma of the skin or any other part of the carcinoma in situ;
7. Have received any other test drug treatment or participated in another interventional clinical trial within 30 days of the screening period;
8. The investigator believes that it is not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 962 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival (DFS) | 3 years
  To evaluate the noninferiority of observation as compared to standard of care adjuvant chemotherapy (investigator's choice) in patients with high-risk stage II CC and High-Immunoscore® in terms of disease free survival (DFS).

SECONDARY OUTCOMES:
Time to Recurrence (TTR) | From date of enrollment until the date of recurrence,assessed 1year,3years and 5years after therapy
  To evaluate the noninferiority of observation as compared to standard of care adjuvant chemotherapy (investigator's choice) in patients with high-risk stage II CC and High-Immunoscore® in terms of Time To Recurrence (TTR)
Overall Survival (OS) | From date of enrollment until the date of death,assessed 1year,3years and 5years after therapy
  To evaluate the noninferiority of observation as compared to standard of care adjuvant chemotherapy (investigator's choice) in patients with high-risk stage II CC and High-Immunoscore® in terms of overall survival (OS)

OTHER OUTCOMES:
Cost Utility Analysis | through study completion,an average of 3 years
  An cost utility analysis at the country level will be conducted alongside the clinical evaluation (exploratory)

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Galon J, Costes A, Sanchez-Cabo F, Kirilovsky A, Mlecnik B, Lagorce-Pages C, Tosolini M, Camus M, Berger A, Wind P, Zinzindohoue F, Bruneval P, Cugnenc PH, Trajanoski Z, Fridman WH, Pages F. Type, density, and location of immune cells within human colorectal tumors predict clinical outcome. Science. 2006 Sep 29;313(5795):1960-4. doi: 10.1126/science.1129139. PMID 17008531
- [Background] Pages F, Kirilovsky A, Mlecnik B, Asslaber M, Tosolini M, Bindea G, Lagorce C, Wind P, Marliot F, Bruneval P, Zatloukal K, Trajanoski Z, Berger A, Fridman WH, Galon J. In situ cytotoxic and memory T cells predict outcome in patients with early-stage colorectal cancer. J Clin Oncol. 2009 Dec 10;27(35):5944-51. doi: 10.1200/JCO.2008.19.6147. Epub 2009 Oct 26. PMID 19858404
- [Background] Mlecnik B, Tosolini M, Kirilovsky A, Berger A, Bindea G, Meatchi T, Bruneval P, Trajanoski Z, Fridman WH, Pages F, Galon J. Histopathologic-based prognostic factors of colorectal cancers are associated with the state of the local immune reaction. J Clin Oncol. 2011 Feb 20;29(6):610-8. doi: 10.1200/JCO.2010.30.5425. Epub 2011 Jan 18. PMID 21245428
- [Background] Mlecnik B, Bindea G, Kirilovsky A, Angell HK, Obenauf AC, Tosolini M, Church SE, Maby P, Vasaturo A, Angelova M, Fredriksen T, Mauger S, Waldner M, Berger A, Speicher MR, Pages F, Valge-Archer V, Galon J. The tumor microenvironment and Immunoscore are critical determinants of dissemination to distant metastasis. Sci Transl Med. 2016 Feb 24;8(327):327ra26. doi: 10.1126/scitranslmed.aad6352. PMID 26912905
- [Background] Mlecnik B, Bindea G, Angell HK, Maby P, Angelova M, Tougeron D, Church SE, Lafontaine L, Fischer M, Fredriksen T, Sasso M, Bilocq AM, Kirilovsky A, Obenauf AC, Hamieh M, Berger A, Bruneval P, Tuech JJ, Sabourin JC, Le Pessot F, Mauillon J, Rafii A, Laurent-Puig P, Speicher MR, Trajanoski Z, Michel P, Sesboue R, Frebourg T, Pages F, Valge-Archer V, Latouche JB, Galon J. Integrative Analyses of Colorectal Cancer Show Immunoscore Is a Stronger Predictor of Patient Survival Than Microsatellite Instability. Immunity. 2016 Mar 15;44(3):698-711. doi: 10.1016/j.immuni.2016.02.025. PMID 26982367
- [Background] Pages F, Mlecnik B, Marliot F, Bindea G, Ou FS, Bifulco C, Lugli A, Zlobec I, Rau TT, Berger MD, Nagtegaal ID, Vink-Borger E, Hartmann A, Geppert C, Kolwelter J, Merkel S, Grutzmann R, Van den Eynde M, Jouret-Mourin A, Kartheuser A, Leonard D, Remue C, Wang JY, Bavi P, Roehrl MHA, Ohashi PS, Nguyen LT, Han S, MacGregor HL, Hafezi-Bakhtiari S, Wouters BG, Masucci GV, Andersson EK, Zavadova E, Vocka M, Spacek J, Petruzelka L, Konopasek B, Dundr P, Skalova H, Nemejcova K, Botti G, Tatangelo F, Delrio P, Ciliberto G, Maio M, Laghi L, Grizzi F, Fredriksen T, Buttard B, Angelova M, Vasaturo A, Maby P, Church SE, Angell HK, Lafontaine L, Bruni D, El Sissy C, Haicheur N, Kirilovsky A, Berger A, Lagorce C, Meyers JP, Paustian C, Feng Z, Ballesteros-Merino C, Dijkstra J, van de Water C, van Lent-van Vliet S, Knijn N, Musina AM, Scripcariu DV, Popivanova B, Xu M, Fujita T, Hazama S, Suzuki N, Nagano H, Okuno K, Torigoe T, Sato N, Furuhata T, Takemasa I, Itoh K, Patel PS, Vora HH, Shah B, Patel JB, Rajvik KN, Pandya SJ, Shukla SN, Wang Y, Zhang G, Kawakami Y, Marincola FM, Ascierto PA, Sargent DJ, Fox BA, Galon J. International validation of the consensus Immunoscore for the classification of colon cancer: a prognostic and accuracy study. Lancet. 2018 May 26;391(10135):2128-2139. doi: 10.1016/S0140-6736(18)30789-X. Epub 2018 May 10. PMID 29754777
- [Background] Sinicrope F et al. Immunoscore to provide prognostic information in low- (T1-3N1) and high-risk (T4 or N2) subsets of stage III colon carcinoma patients treated with adjuvant FOLFOX in a phase III trial (NCCTG N0147; Alliance). J Clin Oncol 36, 2018 (suppl 4S; abstr 614)
- [Background] Galon J, Hermitte F, Mlecnik B, et al. Immunoscore clinical utility to identify good prognostic colon cancer stage II patients with high-risk clinico-pathological features for whom adjuvant treatment may be avoided. J Clin Oncol. 2019;37(4):S487.
- [Background] Pages F, Andre T, Taieb J, et al. Validation of the Immunoscore prognostic value in stage III colon cancer patients treated with oxaliplatin in the prospective IDEA France cohort study (PRODIGE-GERCOR). J Clin Oncol. 2019;37(15):S3513.